CLINICAL TRIAL: NCT03041701
Title: A Phase I/II Trial of the Insulin-Like Growth Factor 1 Receptor (IGF-1R) Antibody AMG479 (Ganitumab) in Combination With the Src Family Kinase (SFK) Inhibitor Dasatinib in Patients With Embryonal and Alveolar Rhabdomyosarcoma
Brief Title: Insulin-like Growth Factor 1 Receptor (IGF-1R) Antibody AMG479 (Ganitumab) in Combination With the Src Family Kinase (SFK) Inhibitor Dasatinib in People With Embryonal and Alveolar Rhabdomyosarcoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The pharmaceutical company discontinued availability of the drug and we were forced to close the study before phase II was completed. Only one participant was enrolled on phase II.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christine Heske, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 170049; 17-C-0049
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Results first posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-03

CONDITIONS: Rhabdomyosarcoma; Rhabdomyosarcoma, Alveolar; Rhabdomyosarcoma, Embryonal
Keywords: ERMS; ARMS; Monoclonal Antibody; YES; RMS
MeSH Terms: conditions — Rhabdomyosarcoma; Rhabdomyosarcoma, Alveolar; Rhabdomyosarcoma, Embryonal | interventions — Dasatinib; ganitumab; Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 Dose Level 1: Ganitumab and Dasatinib (Experimental): Phase I Dose Level 1: Combination of ganitumab and dasatinib with limited dose escalation of dasatinib
  Interventions: Drug: Dasatinib; Drug: Ganitumab
- Phase 1 Dose Level 2: Ganitumab and Dasatinib (Experimental): Phase I Dose Level 2: Combination of ganitumab and dasatinib with limited dose escalation of dasatinib
  Interventions: Drug: Dasatinib; Drug: Ganitumab
- Phase 2 Dose Level 1: Ganitumab and Dasatinib (Experimental): Phase 2 Dose Level 1: Combination of ganitumab and dasatinib at the maximum tolerated dose (MTD) (or highest safe dose)
  Interventions: Drug: Dasatinib; Drug: Ganitumab

INTERVENTIONS:
Drug: Dasatinib — Once daily on days -7 through day 27 during cycle 1, and then days 0-27 for subsequent cycles.
  Other Names: Sprycel
  Arms: Phase 1 Dose Level 1: Ganitumab and Dasatinib; Phase 2 Dose Level 1: Ganitumab and Dasatinib
Drug: Dasatinib — Twice daily on days -7 through day 27 during cycle 1, and then days 0-27 for subsequent cycles.
  Other Names: Sprycel
  Arms: Phase 1 Dose Level 2: Ganitumab and Dasatinib
Drug: Ganitumab — Once every 2 weeks beginning on day 0.
  Other Names: Insulin-like Growth Factor 1 Receptor (IGF-1R) Antibody AMG479

SUMMARY:
Background:

Rhabdomyosarcoma (RMS) is the most common soft tissue sarcoma of childhood. Two types are embryonal RMS (ERMS) and alveolar RMS (ARMS). Dasatinib may block over-expression of a certain enzyme. Ganitumab may block a certain growth factor, which might suppress tumor growth. This drug combination may help slow tumor growth in people with ERMS and ARMS.

Objective:

To see if dasatinib combined with ganitumab is safe and shrinks or slows the growth of tumors in people with ERMS and ARMS.

Eligibility:

People any age who have ERMS or ARMS that did not respond to previous treatment and who can swallow tablets

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Blood, urine, and heart tests
* Scans/x-rays
* Tissue sample: This can be from previous surgery or biopsy.
* Optional biopsy: A small piece of the tumor is removed with a needle.

Participants will be asked to co-enroll in another protocol.

Participants will get a drug interaction handout and wallet card that show what foods and medications to avoid.

Participants will be treated in cycles. The first cycle is 35 days, and the rest are 28 days. Participants will take dasatinib by mouth daily. They will get ganitumab through an intravenous (IV) every 2 weeks. They will have a physical exam every 1-2 weeks, and urine and heart tests before most cycles.

Participants will continue treatment as long as they do not have severe side effects, or their tumors do not get worse.

After ending treatment, participants will have a visit. This includes repeats of the screening tests.

DETAILED DESCRIPTION:
Background:

* Rhabdomyosarcoma (RMS) is the most common soft tissue sarcoma of childhood. The annual incidence in the United States is 4-7 cases per million children under 15 years, which represents 250 new cases per year. Two major histologic subtypes exist: embryonal rhabdomyosarcoma (ERMS) and alveolar rhabdomyosarcoma (ARMS), the latter of which carries a particularly poor prognosis.
* Over-expression of both the type like growth factor 1 (1 IGF) receptor insulin-like growth factor type 1 receptor (IGF-1R) and its ligands has been observed in multiple malignancies, including pediatric sarcomas, and abnormal activation of this pathway contributes to sarcoma development and progression. Downstream signaling cascades of IGF-1R further regulate tumor cell proliferation, survival, and metastasis through the mitogen-activated protein kinase (MAPK)/extracellular signal-regulated kinase 1/2 (ERK) and phosphatidylinositol 3-kinases (PI3Ks)/mammalian target of rapamycin (mTOR) pathways. In the majority of RMS, IGF-1R is highly expressed.
* Monoclonal antibodies targeting IGF-1R interfere with ligand binding and decrease the expression of the receptor on cell surfaces by internalization and degradation of the receptor. A number of these have been tested in the clinical setting. Results from a phase II trial using monotherapy with monoclonal antibodies against IGF-1R resulted in clinically meaningful responses in about 10-15% of patients with RMS. However, the vast majority of these responses were short-lived with a rapid onset of resistance.
* YES is a member of the SRC family tyrosine kinases (SFKs), non-receptor tyrosine kinases that function in a number of signaling pathways necessary for cell growth, differentiation and survival. Preclinical work suggests involvement of YES in a number of solid tumor types, including colon carcinoma, oral squamous cell carcinoma, glioma, pancreatic cancer, mesothelioma, and RMS.
* Recently, the Helman lab published preclinical work showing that in both embryonal and alveolar RMS models, blockade of IGF-1R results in YES activation and that YES activation is associated with resistance to IGF-1R blockade. In addition, combination blockade of IGF-1R and YES in vitro results in downregulation of phospho-AKT in some cell lines. Treatment blocking both IGF-1R and YES results in enhanced growth inhibition of multiple cell lines of both embryonal and alveolar RMS in vitro and in vivo.

Objectives:

1. Phase I: To determine the safe dose of dasatinib when given with ganitumab in patients with relapsed or refractory embryonal or alveolar RMS.
2. Phase II: To determine if the use of ganitumab plus dasatinib is able to be associated with a modest fraction of patients who experience an objective clinical response (complete response (CR) and partial response (PR) as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria. In addition, a second primary objective will estimate the fraction that is without progression at 4 months.

Eligibility:

* Patients must have a diagnosis of relapsed or refractory embryonal or alveolar RMS, be able to swallow tablets, have archival tissue available.
* Patients must have adequate performance status and adequate major organ function and have recovered from acute toxicity of all prior therapies.

Design:

* This is an open label, multi-site, phase I/II study designed to determine if ganitumab given in combination with dasatinib in children and adults with relapsed or refractory embryonal or alveolar RMS for whom no curative options exist.
* In the phase I portion, using a standard 3 + 3 design, limited dose escalations will be performed to define the maximum tolerated dose (MTD) or the highest safe dose tested of dasatinib when given in combination with ganitumab in this patient population.
* In the phase II component, sixteen (16) evaluable patients, including up to 6 patients from the phase I portion treated at the selected phase II dose, will be enrolled to rule out a 5% fraction with a clinical response in favor of a 30% fraction with a clinical response, using a one sided 0.10 significance level exact test for a binomial proportion. In practice, the fraction of the 16 patients that have objective responses will be determined and reported along with 80% and 95% confidence intervals. If there are 3 objective responses in 16 evaluable patients, the lower one-sided exact 90% confidence interval is 7.1%, thus ruling out 5%.
* It is anticipated that approximately 10-15 patients per year may be accrued onto this trial. Thus, 2 to 3 years is expected to completed accrual.
* In all patients, mechanisms of response and resistance will be assessed by analyzing archival tissue for expression of IGF-1R, insulin receptor, IGF-2 expression and phospho-YES expression, and through genomic sequencing (on protocol 10-C-0086). Genomic sequencing of tumor cells from tissue relative to non-tumor cells from whole blood will be profiled to identify the genomic variances that may contribute to response or disease progression and provide an understanding of molecular abnormalities. Ribonucleic acid (RNA) sequencing will be conducted to provide expression data and give relevance to deoxyribonucleic acid (DNA) mutations; Quantitative proteomics analysis will be conducted on all patients to determine the exact amounts of specific proteins and/or to confirm expression of genes that are correlative of response and disease progression. Genomic and transcriptomic analysis will be conducted on patients who consent to protocol 10-C-0086, Comprehensive Omics Analysis of Pediatric Solid Tumors and Establishment of a Repository for Related Biological Studies. All genomic, transcriptomic, and proteomic molecular analyses will be retrospective and exploratory.
* In patients who agree to undergo biopsy of their tumor, provided the tissue is easily accessible and can be biopsied safely with minimal morbidity, mechanisms of response and resistance will be assessed by analyzing biopsy tissue expression of IGF- 1R, insulin receptor, IGF-2 expression and phospho-YES expression, and through genomic sequencing.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients of any age must have histologically or cytologically confirmed embryonal or alveolar rhabdomyosarcoma (RMS) confirmed by the Laboratory of Pathology, National Cancer Institute (NCI) or by the Department of Pathology and Laboratory Medicine, Children's Hospital Los Angeles (CHLA).
* Patients must have measurable disease.
* Patients must be able to undergo appropriate imaging studies to monitor tumor response.
* Archival tissue of tumors (slides or blocks (blocks preferred)) must be available for analysis. If tissue is not available, patients willing to undergo a pre-treatment biopsy may enroll.
* Prior Therapies:

  * There is no maximum number of prior medical therapies.
  * There must be no curative or life prolonging treatments available.
  * Patients who have received other insulin-like growth factor 1 receptor (IGF-1R) antibodies or inhibitors are eligible, as long as an appropriate washout period has elapsed (see below).
  * Participants must have had their last fraction of external beam radiation therapy that is local and palliative at least 2 weeks prior to enrollment (except for radiation therapy to the lungs as noted below) and had their last substantial bone marrow radiation at least 6 weeks prior to enrollment.
  * Participants must have had their last radiation therapy of the lungs at least 8 weeks prior to enrollment.
  * Participants must have had their last dose of temozolomide at least 4 weeks prior to enrollment; their last dose of other cytotoxic chemotherapy at least 3 weeks prior to enrollment; their last dose of biological therapy, such as biological response modifiers (e.g., cytokines), immunomodulatory agents, vaccines, differentiating agents, used to treat their cancer at least 7 days prior to enrollment, their last dose of a monoclonal antibody the shorter of 3 half- lives or 28 days prior to enrollment, and their last dose of any investigational agent at least 4 weeks prior to enrollment.
  * Participants must have recovered from the acute toxic effects of prior therapy to a grade 1 (Common Terminology Criteria for Adverse Events (CTCAE) v.5.0) level prior to enrollment (does not apply to alopecia).
* Age. There are no age limits for this study, but patients must have the ability to swallow tablets.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 or Karnofsky >50% (if greater than or equal to 16 years of age); or children < 16 years old must have a Lansky performance of greater than or equal to 50%.
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count greater than or equal to 1,000/mcL
  * platelets greater than or equal to 75,000/mcL
  * total bilirubin less than or equal to 1.5X upper limit of normal (ULN), with exception of patients with Gilbert syndrome
  * Alanine aminotransferase (ALT) less than or equal to 3.0X upper limit of normal (ULN)
  * creatinine within normal institutional limits OR creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.
  * Normal blood glucose for age
* Hematologic parameters for patients undergoing biopsy only: Patients should have INR less than or equal to 1.4 and prothrombin time (PT) less than or equal to 40 seconds (unless due to lupus anticoagulant). In patients not meeting these parameters, clearance by hematology will be required prior to undergoing a biopsy.
* Cardiac Function: corrected Q-T interval (QTc) < 480 msec, and ejection fraction greater than or equal to 50%
* Contraception. The effects of these agents on the developing human fetus are unknown. For this reason, men and women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 months after completion of administration of either agent. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Negative pregnancy test is required for women of childbearing potential.
* Ability of subject or Legally Authorized Representative (LAR)) to understand and the willingness to sign a written informed consent document.
* Patients will be strongly encouraged to participate in 10-C-0086. If a patient does not agree to enroll on 10-C-0086, germline genetic analysis will not be performed.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dasatinib or ganitumab or other agents used in study.
* Patients who require concurrent treatment with any medications or substances that are potent inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated list, or medical reference text such as the Physician's Desk Reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Patients who require concurrent treatment with antithrombotic and/or anti-platelet agents (e.g., warfarin, heparin, low molecular weight heparin, aspirin, and/or ibuprofen).
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation r surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain dasatinib tablets are excluded.
* Patients with a history of radiation pneumonitis.
* Patients may not have any clinically significant cardiovascular disease including the following:

  * myocardial infarction or ventricular tachyarrhythmia within 6 months
  * major conduction abnormality (unless a cardiac pacemaker is present).

Patients with any cardiopulmonary symptoms of unknown cause (e.g., shortness of breath, chest pain, etc.) should be evaluated by a baseline echocardiogram with or without stress test as needed in addition to electrocardiogram (EKG) to rule out QTc prolongation. The patient may be referred to a cardiologist at the discretion of the principal investigator. Patients with underlying cardiopulmonary dysfunction should be excluded from the study.

* Uncontrolled intercurrent illness including, but not limited to, the following: ongoing or active infection; history of significant bleeding disorder, including congenital (von Willebrands disease) or acquired (anti-factor VIII antibodies) disorders; large pleural effusions; or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with known pre-existing diabetes mellitus will be excluded because of the risk of hyperglycemia with ganitumab.
* Pregnant women are excluded from this study because animal studies with dasatinib have shown embryolethality and fetal skeletal alterations at non-toxic maternal doses. Because there is an unknown but potential risk for adverse events in nursing human infants secondary to treatment of the mother with dasatinib, breastfeeding should be discontinued if the mother is treated with dasatinib.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Heske, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Clinical data available during the study and indefinitely.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be made available via subscription to the Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).
Access Criteria: Clinical data will be made available via subscription to the Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Requests for all collected individual participant data (IPD) data from clinical trials, conducted under a binding collaborative agreement between National Cancer Institute (NCI)/Division of Cancer Treatment and Diagnosis (DCTD) and a pharmaceutical/biotechnology company, that are not under data safety monitoring board (DSMB) monitoring must be in compliance with the terms of the binding collaborative agreement and must be approved by NCI/DCTD and the Pharmaceutical Collaborator (i.e., the NCI Experimental Therapeutics Clinical Trials Network (ETCTN) Director in conjunction with the NCI/DCTD Regulatory Affairs Branch).

REFERENCES:
- [Derived] Akshintala S, Sundby RT, Bernstein D, Glod JW, Kaplan RN, Yohe ME, Gross AM, Derdak J, Lei H, Pan A, Dombi E, Palacio-Yance I, Herrera KR, Miettinen MM, Chen HX, Steinberg SM, Helman LJ, Mascarenhas L, Widemann BC, Navid F, Shern JF, Heske CM. Phase I trial of Ganitumab plus Dasatinib to Cotarget the Insulin-Like Growth Factor 1 Receptor and Src Family Kinase YES in Rhabdomyosarcoma. Clin Cancer Res. 2023 Sep 1;29(17):3329-3339. doi: 10.1158/1078-0432.CCR-23-0709. PMID 37398992
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0049.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Dose Level 1 Dose Escalation Dasatinib 60 mg/m^2 Every Day (QD)/Ganitumab 18 mg/kg: Phase 1 Dose Level 1 Dose Escalation: Dasatinib 60mg/m^2 by mouth (PO) every day (QD) at Day-7. Ganitumab 18mg/kg intravenous (IV) every two weeks starting at Day 0.
  Cycle 1 is Day -7 to 27; all other cycles are Day 0 to 27
- Phase 1 Dose Level 2 Dose Escalation Dasatinib 60 mg/m^2 Twice Daily (BID)/Ganitumab 18 mg/kg: Phase 1 Dose Level 2 Dose Escalation: Dasatinib 60mg/m^2 by mouth (PO) twice a day (BID) at Day-7. Ganitumab 18mg/kg intravenous (IV) every two weeks starting at Day 0.
  Cycle 1 is Day -7 to 27; all other cycles are Day 0 to 27
- Phase 2 Dose Level 1 Maximum Tolerated Dose Dasatinib 60 mg/m^2 Every Day (QD)/ Ganitumab 18 mg/kg: Phase 2 Dose Level 1 Maximum Tolerated Dose: Dasatinib 60mg/m^2 by mouth (PO) every day (QD) at Day-7. Ganitumab 18mg/kg intravenous (IV) every two weeks starting at Day 0.
  Cycle 1 is Day -7 to 27; all other cycles are Day 0 to 27
Period: Ph I: Dose Level 1 and 2 Dose Escalation
Arm/Group | Phase 1 Dose Level 1 Dose Escalation Dasatinib 60 mg/m^2 Every Day (QD)/Ganitumab 18 mg/kg | Phase 1 Dose Level 2 Dose Escalation Dasatinib 60 mg/m^2 Twice Daily (BID)/Ganitumab 18 mg/kg | Phase 2 Dose Level 1 Maximum Tolerated Dose Dasatinib 60 mg/m^2 Every Day (QD)/ Ganitumab 18 mg/kg
Started | 7 | 6 | 0
Completed | 6 | 5 | 0
Not Completed | 1 | 1 | 0
Not completed — Not evaluable for toxicity | 1 | 1 | 0
Period: Ph 2:Dose Level 1 Maximum Tolerated Dose
Arm/Group | Phase 1 Dose Level 1 Dose Escalation Dasatinib 60 mg/m^2 Every Day (QD)/Ganitumab 18 mg/kg | Phase 1 Dose Level 2 Dose Escalation Dasatinib 60 mg/m^2 Twice Daily (BID)/Ganitumab 18 mg/kg | Phase 2 Dose Level 1 Maximum Tolerated Dose Dasatinib 60 mg/m^2 Every Day (QD)/ Ganitumab 18 mg/kg
Started | 0 | 0 | 1
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 1
Not completed — Unacceptable further treatment | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Level 1 Dose Escalation Dasatinib 60 mg/m^2 Every Day (QD)/Ganitumab 18 mg/kg | Phase 1 Dose Level 2 Dose Escalation Dasatinib 60 mg/m^2 Twice Daily (BID)/Ganitumab 18 mg/kg | Phase 2 Dose Level 1 Maximum Tolerated Dose Dasatinib 60 mg/m^2 Every Day (QD)/ Ganitumab 18 mg/kg | Total
Number analyzed (Participants) | 7 | 6 | 1 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 2 | 1 | 7
  Between 18 and 65 years | 3 | 4 | 0 | 7
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.71 (5.15) | 20.17 (8.18) | 5 (0) | 15.86 (7.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 0 | 7
  Male | 1 | 5 | 1 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 0 | 1 | 0 | 1
  Not Hispanic | 5 | 4 | 1 | 10
  Ethnicity unknown | 2 | 1 | 0 | 3
  Black | 0 | 1 | 0 | 1
  White | 6 | 2 | 1 | 9
  Asian | 0 | 2 | 0 | 2
  Race unknown | 0 | 0 | 0 | 0
  White + Unknown | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Safe Dose of Dasatinib When Given With Ganitumab in Participants With Relapsed or Refractory Embryonal or Alveolar Rhabdomyosarcoma (RMS)
Description: The safe dose or maximum tolerated dose (MTD) is defined as the dose level at which no more than 1 of up to 3-6 participants experience a dose-limiting toxicity (DLT) during the first cycle of treatment, and the dose below that at which at least 2 (of ≤6) participants have DLT as a result of the drug. A DLT is any toxicity of grade 3 or higher, with the specific exception of grade 3 nausea and vomiting of < 5 days duration, grade 3 fever or infection < 5 days duration, and grade 3 neutropenia or thrombocytopenia, for example.
Time Frame: First 35 days of treatment
Population: Dasatinib MTD schedule is daily.
Measure: Number; unit: mg/m^2
Groups:
- All Participants: All participants on: Phase 1 Dose Level 1 and Phase 1 Dose Level 2.
Arm/Group | All Participants
Number analyzed (Participants) | 13
mg/m^2 | 60

2. Primary Outcome: Phase II: Number of Participants Who Experience an Objective Clinical Response (CR or PR) When Treated With Ganitumab Plus Dasatinib
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Participants were followed for the duration of their treatment which ranged from 0-6 cycles (each cycle is 28 days) and averaged approximately 2 months.
Population: Per protocol, participants (pts) who receive dasatinib at the maximum tolerated (MTD) dose+ganitumab during phase(ph) I will be included in the evaluation of ph II objectives, if evaluable. 5/7 pts on the Ph 1 at the MTD are evaluable and were analyzed with RECIST (versus 0/7 analyzed) since all evaluable pts underwent disease response analysis. Same applies to ph 2 (1/1 evaluable/analyzed). Pts treated at dose level 2 were not analyzed for this objective because dose level 2 was not the MTD.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Level 1 Dose Escalation Dasatinib 60 mg/m^2 Every Day (QD)/Ganitumab 18 mg/kg | Phase 2 Dose Level 1 Maximum Tolerated Dose Dasatinib 60 mg/m^2 Every Day (QD)/ Ganitumab 18 mg/kg
Number analyzed (Participants) | 5 | 1
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0

3. Primary Outcome: Phase II: Number of Participants That is Without Progression at 4 Months
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Progressive disease is least a 20% increase in the sum of the diameters of target lesions) taking as reference the smallest sum of diameters while on study.
Time Frame: At 4 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Level 1 Dose Escalation Dasatinib 60 mg/m^2 Every Day (QD)/Ganitumab 18 mg/kg | Phase 2 Dose Level 1 Maximum Tolerated Dose Dasatinib 60 mg/m^2 Every Day (QD)/ Ganitumab 18 mg/kg
Number analyzed (Participants) | 5 | 1
Participants | 1 | 0

4. Secondary Outcome: Phase II: Progression Free Survival (PFS) in Participants Receiving Insulin-like Growth Factor 1 Receptor (IGF-1R) Antibody AMG479 (Ganitumab) in Combination With the Src Family Kinase (SFK) Inhibitor Dasatinib
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Progressive disease is at least a 20% increase in the sum of the diameters of target lesions) taking as reference the smallest sum of diameters while on study.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 1 Dose Level 1 Dose Escalation Dasatinib 60 mg/m^2 Every Day (QD)/Ganitumab 18 mg/kg | Phase 2 Dose Level 1 Maximum Tolerated Dose Dasatinib 60 mg/m^2 Every Day (QD)/ Ganitumab 18 mg/kg
Number analyzed (Participants) | 5 | 1
Months | 1.93 [1.67 to 5.83] | 0.88 [NA to NA] — Full range cannot be determined for one participant.

5. Secondary Outcome: Phase II: Number of Participants With Stable Disease >= 6 Months as Defined by the Response Evaluation Criteria in Solid Tumors (RECIST) in Participants Receiving Ganitumab With Dasatinib
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Stable disease is neither sufficient shrinkage to qualify for partial response (i.e., at least a 30% decrease in the sum of the diameters of target lesions) nor sufficient increase to qualify for progressive disease (i.e., at least a 20% increase in the sum of the diameters of target lesions) taking as reference the smallest sum of diameters while on study.
Time Frame: 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Level 1 Dose Escalation Dasatinib 60 mg/m^2 Every Day (QD)/Ganitumab 18 mg/kg | Phase 2 Dose Level 1 Maximum Tolerated Dose Dasatinib 60 mg/m^2 Every Day (QD)/ Ganitumab 18 mg/kg
Number analyzed (Participants) | 5 | 1
Participants | 1 | 0

6. Secondary Outcome: Phase I: Number of Participants With Grade ≥3 Adverse Events Related to Treatment With Ganitumab and Dasatinib
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: Date treatment consent signed to date off study, approximately 14 months and 18 days for phase 1 dose level 1, 27 months and 2 days for phase 1 dose level 2, and 1 month and 24 days for phase 2 dose level 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Level 1 Dose Escalation Dasatinib 60 mg/m^2 Every Day (QD)/Ganitumab 18 mg/kg | Phase 1 Dose Level 2 Dose Escalation Dasatinib 60 mg/m^2 Twice Daily (BID)/Ganitumab 18 mg/kg
Number analyzed (Participants) | 7 | 6
Participants
  Grade 3 related to ganitumab | 1 | 3
  Grade 4 related to ganitumab | 0 | 0
  Grade 5 related to ganitumab | 0 | 0
  Grade 3 related to dasatinib | 3 | 4
  Grade 4 related to dasatinib | 1 | 0
  Grade 5 related to dasatinib | 0 | 0

7. Secondary Outcome: Phase II: Number of Participants With Grade ≥3 Adverse Events Related to Treatment With Ganitumab and Dasatinib
Description: as for outcome 6
Time Frame: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Dose Level 1 Maximum Tolerated Dose Dasatinib 60 mg/m^2 Every Day (QD)/ Ganitumab 18 mg/kg
Number analyzed (Participants) | 1
Participants
  Grade 3 related to ganitumab | 0
  Grade 4 related to ganitumab | 0
  Grade 5 related to ganitumab | 0
  Grade 3 related to dasatinib | 0
  Grade 4 related to dasatinib | 0
  Grade 5 related to dasatinib | 0

8. Other Pre Specified Outcome: Phase I: Number of Participants With a Dose-Limiting Toxicity (DLT)
Description: A DLT is any toxicity of grade 3 or higher, with the specific exception of grade 3 nausea and vomiting of < 5 days duration, grade 3 fever or infection < 5 days duration, and grade 3 neutropenia or thrombocytopenia, for example.
Time Frame: First 35 days of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Level 1 Dose Escalation Dasatinib 60 mg/m^2 Every Day (QD)/Ganitumab 18 mg/kg | Phase 1 Dose Level 2 Dose Escalation Dasatinib 60 mg/m^2 Twice Daily (BID)/Ganitumab 18 mg/kg
Number analyzed (Participants) | 7 | 6
Participants | 1 | 2

9. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Level 1 Dose Escalation Dasatinib 60 mg/m^2 Every Day (QD)/Ganitumab 18 mg/kg | Phase 1 Dose Level 2 Dose Escalation Dasatinib 60 mg/m^2 Twice Daily (BID)/Ganitumab 18 mg/kg | Phase 2 Dose Level 1 Maximum Tolerated Dose Dasatinib 60 mg/m^2 Every Day (QD)/ Ganitumab 18 mg/kg
Number analyzed (Participants) | 7 | 6 | 1
Participants | 7 | 6 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 14 months and 18 days for phase 1 dose level 1, 27 months and 2 days for phase 1 dose level 2, and 1 month and 24 days for phase 2 dose level 1.
Arm/Group | Phase 1 Dose Level 1 Dose Escalation Dasatinib 60 mg/m^2 Every Day (QD)/Ganitumab 18 mg/kg | Phase 1 Dose Level 2 Dose Escalation Dasatinib 60 mg/m^2 Twice Daily (BID)/Ganitumab 18 mg/kg | Phase 2 Dose Level 1 Maximum Tolerated Dose Dasatinib 60 mg/m^2 Every Day (QD)/ Ganitumab 18 mg/kg
All-Cause Mortality (participants affected / at risk) | 2/7 | 1/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 4/7 | 5/6 | 1/1
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1 Dose Escalation Dasatinib 60 mg/m^2 Every Day (QD)/Ganitumab 18 mg/kg (N=7) | Phase 1 Dose Level 2 Dose Escalation Dasatinib 60 mg/m^2 Twice Daily (BID)/Ganitumab 18 mg/kg (N=6) | Phase 2 Dose Level 1 Maximum Tolerated Dose Dasatinib 60 mg/m^2 Every Day (QD)/ Ganitumab 18 mg/kg (N=1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Infections and infestations - Other, Blood culture positive for Klebsiella pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1 Dose Escalation Dasatinib 60 mg/m^2 Every Day (QD)/Ganitumab 18 mg/kg (N=7) | Phase 1 Dose Level 2 Dose Escalation Dasatinib 60 mg/m^2 Twice Daily (BID)/Ganitumab 18 mg/kg (N=6) | Phase 2 Dose Level 1 Maximum Tolerated Dose Dasatinib 60 mg/m^2 Every Day (QD)/ Ganitumab 18 mg/kg (N=1)
Abdominal distension (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 2 (3) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (6) | 2 (11) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 2 (6) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 7 (31) | 6 (25) | 1 (4)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (10) | 4 (14) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (9) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cardiac troponin T increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (6) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 3 (4) | 0 (0)
Creatinine increased (Investigations) | 1 (2) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (8) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 3 (21) | 0 (0)
Edema face (General disorders) | 1 (1) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 2 (3) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 1 (1)
Eye disorders - Other, Left eye/ medial SCH-Irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (8) | 3 (3) | 0 (0)
Fever (General disorders) | 3 (12) | 3 (14) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Mild tenderness in lower right quadrant (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Gagging (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Lower lip pressure ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Oral bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Oral ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, Difficulty with accessing port (General disorders) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, Specify (General disorders) | 1 (1) | 0 (0) | 0 (0) — Pain associated with nephrostomy tube placement
General disorders and administration site conditions - Other, Superficial edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 2 (3) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (5) | 4 (4) | 0 (0)
Hemoglobinuria (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (6) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (6) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (14) | 5 (16) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (17) | 5 (11) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (9) | 4 (6) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 5 (12) | 5 (9) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (18) | 2 (5) | 0 (0)
Hypotension (Vascular disorders) | 3 (5) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Investigations) | 2 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 5 (15) | 5 (22) | 0 (0)
Lymphocyte count increased (Investigations) | 1 (1) | 2 (3) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, Appetite decrease (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, Appetite slight decrease (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, Decrease in appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Metabolism and nutrition disorders - Other, Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Tenderness to palpation over posterior lower left ribs
Musculoskeletal and connective tissue disorder - Other, Specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Tenderness to palpation right upper back and lateral chest
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (11) | 2 (3) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (7) | 2 (5) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Periorbital edema (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 7 (17) | 6 (12) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 2 (14) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 7 (15) | 4 (9) | 0 (0)
Psychiatric disorders - Other, Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders - Other, Restless legs (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders - Other, Sleep disturbance (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, Mild suprapubic distention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, White blood cell, Urine increased (Renal and urinary disorders) | 2 (5) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, L nasal fullness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Some congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Tachypnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 4 (12) | 2 (3) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Candida diaper rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Diaper rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Erythema/ pressure sore L.buttock (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Insect bites (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, Pain lateral of port access (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tricuspid valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (7) | 2 (2) | 1 (2)
Weight gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 3 (12) | 3 (10) | 1 (2)
General disorders and administration site conditions-Other, pain associated with suprapubic catheter (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT03041701/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT03041701/ICF_001.pdf